CLINICAL TRIAL: NCT00000793
Title: A Phase II/III Double-Blind Study of Amitriptyline and Mexiletine for Painful Neuropathy in HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 242; 11219 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Peripheral Nervous System Disease
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Peripheral Nervous System Diseases; Amitriptyline; Pain; Mexiletine; benzatropine methanesulfonate; Parasympatholytics
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Pain | interventions — Mexiletine; Benztropine; Amitriptyline

INTERVENTIONS:
Drug: Mexiletine hydrochloride
Drug: Benztropine mesylate
Drug: Amitriptyline hydrochloride

SUMMARY:
To assess the efficacy, safety, and tolerability of amitriptyline hydrochloride versus mexiletine hydrochloride in reducing pain intensity in patients with HIV-related painful peripheral neuropathy.

No large-scale controlled clinical trials of symptomatic therapy for painful HIV-related neuropathy have been attempted. Both amitriptyline and mexiletine have been useful in the management of painful neuropathies; however, both are associated with certain toxicities. In this comparative study of amitriptyline and mexiletine, benztropine mesylate also will be included as an active placebo to mimic the side effects of the study drugs.

DETAILED DESCRIPTION:
No large-scale controlled clinical trials of symptomatic therapy for painful HIV-related neuropathy have been attempted. Both amitriptyline and mexiletine have been useful in the management of painful neuropathies; however, both are associated with certain toxicities. In this comparative study of amitriptyline and mexiletine, benztropine mesylate also will be included as an active placebo to mimic the side effects of the study drugs.

Patients are randomized to receive amitriptyline, mexiletine, or benztropine mesylate as an active placebo to mimic the mild side effects associated with both amitriptyline and mexiletine. Doses are gradually increased over 4 weeks until a minimum effective dose or MTD is reached, then patients are treated for at least 4 additional weeks at the final dose before gradually tapering off. Neurologic exams are performed at screening and at the end of treatment. Intensity of pain is rated twice daily by the patient. Patients are followed at Weeks 2, 4, and 8, and at 10 days after completely tapering off of drug.

PER 3/16/95 AMENDMENT: Patients with no pain relief 14 days after initiation of study therapy may have dose doubled or increased to maximum allowable dose, whichever is lower. Then if no improvement occurs within 14 days after dose increase, patients have the option of discontinuing study medication.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aspirin and acetaminophen.
* Nonsteroidal anti-inflammatory agents.
* Opiates.
* Pyridoxine (only if accompanied by isoniazid).
* ddI, ddC, d4T, and 3TC if on a stable dose.
* AZT.
* Cimetidine if on a stable dose.

NOTE:

* Per 3/16/95 amendment, Lactaid may be taken by lactose-intolerant patients for effects of lactose in placebo capsules.

Concurrent Treatment:

Allowed:

* Acupuncture.

Patients must have:

* Documented HIV infection.
* Painful peripheral neuropathy.

NOTE:

* Patients in ACTG blinded studies of dideoxynucleosides such as ddI, ddC, and d4T are encouraged to enroll in this study.

Prior Medication:

Allowed:

* Prior ddI, ddC, d4T, or 3TC, if on a stable dose for at least 8 weeks prior to study entry.
* Prior cimetidine if on a stable dose for at least 2 weeks prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Diabetes mellitus.
* Neurological disease of sufficient severity to confound the evaluation of peripheral neuropathy, such as myelopathy without neuropathy. (NOTE: Patients with both myelopathy AND painful peripheral neuropathy are eligible.)
* Electrocardiogram (EKG) indicating malignant arrhythmia or cardiac conduction disturbances (such as second or third degree AV block, anterior hemi-block, or prolonged QT interval).
* Suicidal thoughts of sufficient severity to require treatment with antidepressant medication.

Concurrent Medication:

Excluded:

* Phenytoin or carbamazepine (unless on stable dose for 8 weeks prior to study entry).
* Capsaicin.
* Any MAO inhibitor antidepressants, any tricyclic or tetracyclic antidepressants, certain serotonin re-uptake inhibitors (fluoxetine, paroxetine, and venlafaxine), or mexiletine (except as dispensed for this study).
* Disopyramide.
* Procainamide.
* Quinidine.
* Tocainide.
* Flecainide acetate.
* Encainide.
* Lidocaine.
* Cisplatin.
* Vincristine.
* Chloramphenicol, disulfiram, ethionamide glutethimide, gold, hydralazine, iodoquinol, metronidazole, nitrofurantoin, or ribavirin (only in patients in whom the onset or clear worsening of painful peripheral neuropathy was attributed to previously taking these drugs).
* Any investigational drugs other than 3TC (except with permission of the protocol team).
* Terfenadine (if concurrent with ketoconazole).

Patients with the following prior conditions are excluded:

* Documented history of cardiac disease.
* History of allergy to, or intolerance of, tricyclic antidepressants, mexiletine, or benztropine.

Prior Medication:

Excluded:

* Prior disopyramide.
* Prior procainamide.
* Prior quinidine.
* Prior tocainide.
* Prior flecainide acetate.
* Prior encainide.
* Prior lidocaine.
* Cisplatin or vincristine within 8 weeks prior to study entry.
* Chloramphenicol, disulfiram, ethionamide glutethimide, gold, hydralazine, iodoquinol, metronidazole, nitrofurantoin, or ribavirin within 8 weeks prior to study entry (only in patients in whom the onset or clear worsening of painful peripheral neuropathy was attributed to taking these drugs).
* Any MAO inhibitor antidepressants, any tricyclic or tetracyclic antidepressants, certain serotonin re-uptake inhibitors (fluoxetine, paroxetine, and venlafaxine), or mexiletine, within 4 weeks prior to study entry.
* More than 50 percent change in the weekly dosage of any pain control medications within 2 weeks prior to study entry.

Per 3/16/95 amendment:

* ddI, ddC, d4T, or 3TC within 8 weeks prior to study entry ONLY IF dideoxynucleoside dosing was suspended or permanently discontinued.

Risk Behavior:

Excluded:

* Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Study Completion 1997-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K Kieburtz, Study Chair; D Simpson, Study Chair
Locations (37):
- United States (36):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Hennepin County Med. Ctr., Div. of Infectious Diseases, Minneapolis, Minnesota
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Lein B. Potential therapy for painful neuropathy. PI Perspect. 1995 May;(no 16):11. PMID 11362419
- [Background] Kieburtz K, Simpson D, Yiannoutsos C, Max MB, Hall CD, Ellis RJ, Marra CM, McKendall R, Singer E, Dal Pan GJ, Clifford DB, Tucker T, Cohen B. A randomized trial of amitriptyline and mexiletine for painful neuropathy in HIV infection. AIDS Clinical Trial Group 242 Protocol Team. Neurology. 1998 Dec;51(6):1682-8. doi: 10.1212/wnl.51.6.1682. PMID 9855523